CLINICAL TRIAL: NCT01341990
Title: Effect of SiH MPDS FID 114675A vs. a Marketed Multi-Purpose Solution on Lens Moisture
Brief Title: Effect of an Investigational Multi-Purpose Solution on Lens Moisture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: C-09-031
Record Dates: First submitted 2009-12-09; First posted 2011-04-26 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-03

CONDITIONS: Contact Lens Moisture
Keywords: Contact Lenses; Contact Lens Care; Multi-Purpose Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 114675A (Experimental): Multi-purpose disinfecting solution used per protocol-specified instructions for cleaning, rinsing, disinfecting/storing, and reinserting study contact lenses
  Interventions: Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS); Device: Silicone Hydrogel Contact Lenses
- ReNu MultiPlus (Active Comparator): Multi-purpose solution used per protocol-specified instructions for cleaning, rinsing, disinfecting/storing, and reinserting study contact lenses
  Interventions: Device: ReNu Fresh Lens Comfort Multi-Purpose Solution (MPS); Device: Silicone Hydrogel Contact Lenses

INTERVENTIONS:
Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS) — Investigational solution intended for use as a cleaning, rinsing, reconditioning, disinfecting, and storage solution for silicone hydrogel and soft contact lenses
  Arms: FID 114675A
Device: ReNu Fresh Lens Comfort Multi-Purpose Solution (MPS) — Commercially marketed prodouct indicated for cleaning, removing protein deposits, rinsing, disinfecting, and storing soft contact lenses
  Other Names: ReNu MultiPlus® Multi-Purpose Solution Fresh Lens Comfort™
  Arms: ReNu MultiPlus
Device: Silicone Hydrogel Contact Lenses — Commercially marketed silicone hydrogel contact lenses per habitual prescription for daily wear use, at least 8 hours/day. New pair dispensed at Day 0 (Baseline Visit) and at the conclusion of Day 1 (Visit 2).
  Other Names: Acuvue® Oasys™; PureVision®

SUMMARY:
The purpose of the study is to evaluate the effect of an investigational multi-purpose disinfecting solution (MPDS) compared to a marketed multi-purpose solution on the moisture of silicone hydrogel contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Wears silicone hydrogel contact lenses on a daily wear basis i.e. disinfects lenses every night).
* Has successfully worn contact lenses for 5 days, 8 hours per day, prior to baseline visit.
* Vision is correctable to 20/30 or better in each eye at distance with study lenses at baseline visit.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Known sensitivity or intolerance to contact lens multi-purpose solutions.
* Use of any topical ocular OTC or prescribed topical ocular medications.
* History or current ocular infections or ocular inflammatory events.
* Ocular surgery within the past year.
* Medical condition or use of medication that cause ocular side effects.
* Participation in any investigational study within the past 30 days.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin R Webb, OD, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 US study center.
Period: Overall Study
Arm/Group | FID 114675A | ReNu MultiPlus
Started | 35 | 33
Completed | 32 | 32
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Torn Study Lens | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FID 114675A | ReNu MultiPlus | Total
Number analyzed (Participants) | 35 | 33 | 68
Age Continuous [Mean (Standard Deviation); unit: years] | 43.9 (9.2) | 42.8 (11.2) | 43.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 35 | 33 | 68

OUTCOME MEASURES:

1. Primary Outcome: Mean Ex-Vivo Advancing Contact Angle
Description: Study lens was removed from the eye according to protocol-specified procedures. The OCA15 (Optical Contact Angle) Instrument was used to observe, record, and calculate contact angle measurements. The wetting angle measurement was recorded in degrees (0-180), and a lower wetting angle measurement indicates a more wettable lens.
Time Frame: Day 1, 8 hours
Population: Intent to Treat.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | FID 114675A | ReNu MultiPlus
Number analyzed (Participants) | 34 | 32
Degrees | 56.7 (21.2) | 59.2 (23.7)

2. Primary Outcome: Mean Ex-Vivo Advancing Contact Angle
Description: as for outcome 1
Time Frame: Day 8, 16 hours
Population: Intent to treat.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | FID 114675A | ReNu MultiPlus
Number analyzed (Participants) | 31 | 32
Degrees | 59.5 (21.2) | 63.4 (17.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 23 Nov 2009 to 27 Jan 2010.
Arm/Group | FID 114675A | ReNu MultiPlus
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes